CLINICAL TRIAL: NCT01527175
Title: Comparision of Ultrasound-guided Supraclavicular and Infraclavicular Approach for Central Venous Catheterization in Children
Brief Title: Ultrasound-guided Subclavian Venous Catheterization in Children
Acronym: SuCVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JNB-KJT-12
Record Dates: First submitted 2012-01-28; First posted 2012-02-06 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Subclavian Venous Catheterization in Children

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- supraclavicular (Active Comparator): supraclavicular: supraclavicular approach for subclavian venous catheterization
  Interventions: Other: Approach for ultrasound-guided subclavian venous catheterization
- infraclavicular (Placebo Comparator): infraclavicular: infraclavicular approach for subclavian venous catheterization
  Interventions: Other: Approach for ultrasound-guided subclavian venous catheterization

INTERVENTIONS:
Other: Approach for ultrasound-guided subclavian venous catheterization — Each SCV catheterization was performed under ultrasound-guidance with supraclvicular or infraclavicular approach.

SUMMARY:
The subclavian vein (SCV) is often the preferred site for central venous access. Ultrasound-guided SCV catheterizations with supraclavicular (SC) or infraclavicular (IC) approach have been proved to be useful in children. The investigators compared the success rate, number of attempts, time tocatheterization, and complication.

ELIGIBILITY:
Inclusion Criteria:

* central venous lines required patients
* children < 10 yr of age

Exclusion Criteria:

* inadequate ultrasound visualization of the subclavian vein

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The duration for susscessful placement of needle into subclavian vein | within 20 minutes
  The time needed to place needle into the vein (from needle entry into the skin to aspiration of blood with syringe) was measured. When the duration was recorded as greater than 20 min, the procedure was defined unsuccessful and excluded from the analysis.

SECONDARY OUTCOMES:
The number of attempt for susscessful placement of needle into subclavian vein. | within 20 minutes
  An 'attempt' was defined as each needle advancement to place needl into the vein. When the duration for susscessful placement of needle into subclavian vein was recorded as greater than 20 min, the procedure was defined unsuccessful and excluded from the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea

REFERENCES:
- [Derived] Byon HJ, Lee GW, Lee JH, Park YH, Kim HS, Kim CS, Kim JT. Comparison between ultrasound-guided supraclavicular and infraclavicular approaches for subclavian venous catheterization in children--a randomized trial. Br J Anaesth. 2013 Nov;111(5):788-92. doi: 10.1093/bja/aet202. Epub 2013 Jun 10. PMID 23756247